CLINICAL TRIAL: NCT00461630
Title: A Randomized Trial of the Long-term Clinical Effects of Raising HDL Cholesterol With Extended Release Niacin/Laropiprant
Brief Title: Treatment of HDL to Reduce the Incidence of Vascular Events HPS2-THRIVE
Acronym: HPS2-THRIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jane Armitage, Professor of Clinical trials and Epidemiology, Clinical trial Service Unit & Epidemiological Studies Unit (CTSU), Nuffield Department of Clinical Medicine, University of Oxford, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTSUTHRIVE1; ISRCTN29503772; 2006-001885-17 (EudraCT Number)
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Cardiovascular Disease; Peripheral Arterial Disease; Diabetes Mellitus; Coronary Heart Disease
Keywords: coronary heart disease; cardiovascular disease; stroke; peripheral arterial disease; diabetes mellitus; cholesterol; HDL cholesterol; simvastatin; ezetimibe; ER niacin; laropiprant
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Arterial Disease; Diabetes Mellitus; Coronary Disease; Stroke | interventions — MK-0524; Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ER niacin/laropiprant (Experimental): 1 g ER niacin plus 20 mg laropiprant per tablet. 2 tablets orally per day. With either 40 mg simvastatin tablet or ezetimibe/simvastatin (10 mg/40 mg) in single tablet taken once daily
  Interventions: Drug: ER niacin/laropiprant; Drug: simvastatin; Drug: ezetimibe/simvastatin
- Placebo (Active Comparator): Placebo (for ER niacin/laropiprant) 2 tablets orally per day. With either 40 mg simvastatin tablet orally per day or ezetimibe/simvastatin (10 mg/40 mg) in single tablet taken once daily
  Interventions: Drug: simvastatin; Drug: ezetimibe/simvastatin

INTERVENTIONS:
Drug: ER niacin/laropiprant
  Other Names: Tredaptive
  Arms: ER niacin/laropiprant
Drug: simvastatin — 40 mg simvastatin tablet orally per day as background LDL-lowering treatment allocated at entry based on previous statin treatment and total cholesterol level
  Other Names: Zocor
Drug: ezetimibe/simvastatin — 10 mg ezetimibe plus 40 mg simvastatin in single tablet taken once daily as background LDL-lowering treatment allocated at entry based on previous statin treatment and total cholesterol level
  Other Names: Inegy; Vytorin

SUMMARY:
The primary aim is to assess the effects of raising HDL cholesterol (the good type) with extended release niacin/laropiprant 2g (previously known as MK-0524A) versus matching placebo on the risk of heart attack or coronary death, stroke, or the need for arterial bypass procedures (revascularisation) in people with a history of circulatory problems. The secondary aim is to assess the effects of extended release niacin/laropiprant 2g daily on heart attack, coronary death, stroke, and revascularisation separately and to assess the effects on mortality both overall and in various categories of causes of death, and of the effects on major cardiovascular events in people with a history of different diseases at the beginning of the study.

DETAILED DESCRIPTION:
Cardiovascular disease is one of the leading causes of morbidity and mortality in the United Kingdom (UK), as well as in the developed and the developing world. Finding new and safe treatments to reduce the burden of heart disease and strokes is therefore an important contribution to public health and in the wider public interest. HPS2-THRIVE aims to find out whether by combining niacin (a drug that has been available for 50 years) with a new drug laropiprant(which reduces the side-effects of niacin) is beneficial. All participants in HPS2-THRIVE will have established cardiovascular disease and therefore be at very high risk of recurrent vascular events (myocardial infarction, stroke or the need for arterial revascularisation). Two of the most important risk factors for recurrent events in such patients are the blood levels of LDL cholesterol with a positive association, and HDL cholesterol levels with a negative association.

HDL cholesterol has long been known to have a strong inverse correlation with coronary heart disease (CHD) risk. But, randomized trial evidence for beneficial effects from raising HDL cholesterol is limited. One of the most effective HDL-raising agents is niacin but the tolerability of niacin has been severely limited by flushing and cutaneous side-effects, which appear to be mediated largely by prostaglandin D. Laropiprant is a selective prostaglandin D receptor antagonist that substantially reduces the frequency and intensity of niacin-induced flushing. Daily oral doses of extended release (ER) niacin plus Laropiprant 2g(formerly MK-0524A) have been well tolerated in early studies and increase HDL cholesterol by 20-25%. The trial will assess whether this increase in HDL cholesterol translates into clinical benefit as is expected from the observational evidence. In addition, all participants will also be provided with effective LDL-lowering therapy, as either simvastatin 40mg daily alone or with ezetimibe 10mg daily in a combination tablet.

The complementary effects on the HDL (good) and LDL (bad) cholesterol produced by extended release niacin/laropiprant 2 g daily and simvastatin 40 mg with or without ezetimibe 10 mg should provide an excellent treatment option for patients with vascular disease. However, no trials so far have demonstrated clearly that raising HDL cholesterol produces the expected reduction in cardiovascular risk. If HPS2-THRIVE is able to demonstrate reliably that raising HDL cholesterol reduces the risk of further cardiovascular events then this will be relevant to hundreds of millions of people worldwide.

ELIGIBILITY:
Inclusion Criteria:

* History of myocardial infarction; or
* Cerebrovascular atherosclerotic disease (history of presumed ischaemic stroke, transient ischaemic attack or carotid revascularisation)
* Peripheral arterial disease (i.e. intermittent claudication or history of revascularisation); or
* Diabetes mellitus with any of the above or with other evidence of symptomatic coronary heart disease (i.e. stable or unstable angina, or a history of coronary revascularisation or acute coronary syndrome).

Exclusion Criteria:

* Age <50 or >80 years at invitation to Screening;
* Less than 3 months since presentation with acute myocardial infarction, coronary syndrome or stroke (but such patients may be entered later, if appropriate);
* Planned revascularisation procedure within 3 months after randomization (but such patients may be entered later, if appropriate);
* Definite history of chronic liver disease, or abnormal liver function (i.e. Alanine transaminase (ALT) >1.5 times upper limit of normal (ULN). (Note: Patients with a history of acute hepatitis are eligible provided this ALT limit is not exceeded);
* Breathlessness at rest for any reason;
* Severe renal insufficiency (i.e. creatinine >200 µmol/L);
* Evidence of active inflammatory muscle disease (e.g. dermatomyositis, polymyositis), or Creatine kinase (CK) >3 times upper limit of normal (3xULN);
* Previous significant adverse reaction to a statin, ezetimibe, niacin or laropiprant;
* Active peptic ulcer disease;
* Concurrent treatment with:
* fibric acid derivative ("fibrate")
* niacin (nicotinic acid) at doses more than 100 mg daily
* ezetimibe in combination with either simvastatin 80 mg, or atorvastatin 20-80 mg, or rosuvastatin 10-40 mg daily
* any potent cytochrome P450 3A4 (CYP3A4) inhibitor, including: macrolide antibiotics (erythromycin, clarithromycin, telithromycin); systemic use of imidazole or triazole antifungals (e.g. itraconazole, ketoconazole); protease inhibitors (antiretroviral drugs for HIV infection); and nefazodone
* ciclosporin
* amiodarone
* verapamil
* danazol (Note: Patients who are temporarily taking such drugs may be re-screened when they discontinue them, if considered appropriate.);
* Known to be poorly compliant with clinic visits or prescribed medication;
* Medical history that might limit the individual's ability to take trial treatments for the duration of the study (e.g. severe respiratory disease, history of cancer or evidence of spread within last 5 years other than non-melanoma skin cancer, or recent history of alcohol or substance misuse)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25673 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Armitage, Principal Investigator — Clinical Trial Service Unit, University of Oxford; Colin Baigent, Principal Investigator — Clinical Trial service Unit, University of Oxford; Zhengming Chen, Principal Investigator — Clinical Trial Service Unit, University of Oxford; Martin Landray, Principal Investigator — Clinical Trial Service Unit, University of Oxford
Locations (1):
- Clinical Trial Service Unit, University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] HPS2-THRIVE Collaborative Group; Haynes R, Chen F, Wincott E, Dayanandan R, Lay MJ, Parish S, Bowman L, Landray MJ, Armitage J. Investigating modifications to participant information materials to improve recruitment into a large randomized trial. Trials. 2019 Dec 5;20(1):681. doi: 10.1186/s13063-019-3779-4. PMID 31805983
- [Derived] Haynes R, Valdes-Marquez E, Hopewell JC, Chen F, Li J, Parish S, Landray MJ, Armitage J; HPS2-THRIVE Collaborative Group; HPS2-THRIVE Writing Committee members; HPS2-THRIVE Steering Committee members. Serious Adverse Effects of Extended-release Niacin/Laropiprant: Results From the Heart Protection Study 2-Treatment of HDL to Reduce the Incidence of Vascular Events (HPS2-THRIVE) Trial. Clin Ther. 2019 Sep;41(9):1767-1777. doi: 10.1016/j.clinthera.2019.06.012. Epub 2019 Aug 22. PMID 31447131
- [Derived] Offer A, Arnold M, Clarke R, Bennett D, Bowman L, Bulbulia R, Haynes R, Li J, Hopewell JC, Landray M, Armitage J, Collins R, Parish S; Heart Protection Study (HPS), Study of the Effectiveness of Additional Reductions in Cholesterol and Homocysteine (SEARCH), and Treatment of HDL (High-Density Lipoprotein) to Reduce the Incidence of Vascular Events (HPS2-THRIVE) Collaborative Grou. Assessment of Vascular Event Prevention and Cognitive Function Among Older Adults With Preexisting Vascular Disease or Diabetes: A Secondary Analysis of 3 Randomized Clinical Trials. JAMA Netw Open. 2019 Mar 1;2(3):e190223. doi: 10.1001/jamanetworkopen.2019.0223. PMID 30821829
- [Derived] Parish S, Hopewell JC, Hill MR, Marcovina S, Valdes-Marquez E, Haynes R, Offer A, Pedersen TR, Baigent C, Collins R, Landray M, Armitage J; HPS2-THRIVE Collaborative Group. Impact of Apolipoprotein(a) Isoform Size on Lipoprotein(a) Lowering in the HPS2-THRIVE Study. Circ Genom Precis Med. 2018 Feb;11(2):e001696. doi: 10.1161/CIRCGEN.117.001696. PMID 29449329
- [Derived] Kent S, Haynes R, Hopewell JC, Parish S, Gray A, Landray MJ, Collins R, Armitage J, Mihaylova B; HPS2-THRIVE Collaborative Group. Effects of Vascular and Nonvascular Adverse Events and of Extended-Release Niacin With Laropiprant on Health and Healthcare Costs. Circ Cardiovasc Qual Outcomes. 2016 Jul;9(4):348-54. doi: 10.1161/CIRCOUTCOMES.115.002592. Epub 2016 Jul 12. PMID 27407053
- [Derived] HPS2-THRIVE Collaborative Group; Landray MJ, Haynes R, Hopewell JC, Parish S, Aung T, Tomson J, Wallendszus K, Craig M, Jiang L, Collins R, Armitage J. Effects of extended-release niacin with laropiprant in high-risk patients. N Engl J Med. 2014 Jul 17;371(3):203-12. doi: 10.1056/NEJMoa1300955. PMID 25014686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 245 sites January 2007 to July 2010
Pre-assignment Details: Prior to randomization, each participant received simvastatin 40mg daily; if this dose was not as effective as their prior statin treatment or their total cholesterol was ≥135 mg/dl after 4 weeks on simvastatin alone, ezetimibe 10mg daily was added. Participants then received ERN/LRPT 1g/20mg daily for 4 weeks followed by 2g/40mg daily for 4 weeks.
Groups:
- ER Niacin/Laropiprant: I g ER niacin plus 20mg laropiprant per tablet. 2 tablets orally per day. With either 40 mg simvastatin tablet or ezetimibe/simvastatin (10 mg/40 mg) in single tablet taken once daily
Period: Overall Study
Arm/Group | ER Niacin/Laropiprant | Placebo
Started | 12838 | 12835
Completed | 11932 | 12008
Not Completed | 906 | 827
Not completed — Death | 798 | 732
Not completed — Lost to Follow-up | 108 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ER Niacin/Laropiprant | Placebo | Total
Number analyzed (Participants) | 12838 | 12835 | 25673
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6470 | 6462 | 12932
  >=65 years | 6368 | 6373 | 12741
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 64.9 (7.5) | 64.9 (7.5) | 64.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2224 | 2220 | 4444
  Male | 10614 | 10615 | 21229
Region of Enrollment [Number; unit: participants]
  China | 5464 | 5468 | 10932
  Europe | 7374 | 7367 | 14741

OUTCOME MEASURES:

1. Primary Outcome: Major Vascular Event
Description: Non-fatal myocardial infarction or coronary death, non-fatal or fatal stroke, or revascularisation
Time Frame: During scheduled treatment period (median duration 3.9 years)
Measure: Number; unit: participants
Arm/Group | ER Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 12838 | 12835
participants | 1696 | 1758

2. Secondary Outcome: Major Coronary Events
Description: Non-fatal myocardial infarction (MI) or coronary death
Time Frame: During scheduled treatment period (median duration 3.9 years)
Measure: Number; unit: participants
Arm/Group | ER Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 12838 | 12835
participants | 668 | 694

3. Secondary Outcome: Stroke
Description: Fatal or non-fatal
Time Frame: During scheduled treatment period (median duration 3.9 years)
Measure: Number; unit: participants
Arm/Group | ER Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 12838 | 12835
participants | 498 | 499

4. Secondary Outcome: Coronary or Non-coronary Revascularisation
Time Frame: During scheduled treatment period (median duration 3.9 years)
Measure: Number; unit: participants
Arm/Group | ER Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 12838 | 12835
participants | 807 | 897

5. Secondary Outcome: Mortality
Description: All-cause mortality
Time Frame: During scheduled treatment period (median duration 3.9 years)
Measure: Number; unit: participants
Arm/Group | ER Niacin/Laropiprant | Placebo
Number analyzed (Participants) | 12838 | 12835
participants | 798 | 732

ADVERSE EVENTS:
Time Frame: Mean 3.6 year follow-up
Description: Adverse Events were analyzed at the System Organ Class (SOC) level. All Serious Adverse Events were recorded, but non-serious adverse events were only recorded if considered by participant to be related to study treatment.
Arm/Group | ER Niacin/Laropiprant | Placebo
Serious Adverse Events (participants affected / at risk) | 7137/12838 | 6762/12835
Other Adverse Events (participants affected / at risk) | 4248/12838 | 2238/12835
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ER Niacin/Laropiprant (N=12838) | Placebo (N=12835)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 84 | 56
Cardiac disorders (Cardiac disorders) | 1937 | 1925
Congenital, familial, genetic disorders (Congenital, familial and genetic disorders) | 28 | 19
Ear and labyrinth disorders (Ear and labyrinth disorders) | 52 | 40
Eye disorders (Eye disorders) | 50 | 75
Gastrointestinal disorders (Gastrointestinal disorders) | 620 | 491
General disorders (General disorders) | 346 | 300
Hepatobiliary disorders (Hepatobiliary disorders) | 163 | 140
Immune system disorders (Immune system disorders) | 20 | 25
Infections and infestations (Infections and infestations) | 1031 | 853
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 456 | 400
Investigations (Investigations) | 1210 | 1108
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 961 | 703
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 446 | 364
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 751 | 749
Nervous system disorders (Nervous system disorders) | 1067 | 1086
Psychiatric disorders (Psychiatric disorders) | 68 | 65
Renal and urinary disorders (Renal and urinary disorders) | 208 | 188
Reproductive system and breast disorders (Reproductive system and breast disorders) | 41 | 40
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 358 | 307
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 86 | 51
Social circumstances (Social circumstances) | 0 | 1
Surgical and medical procedures (Surgical and medical procedures) | 2721 | 2722
Vascular disorders (Vascular disorders) | 258 | 246
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ER Niacin/Laropiprant (N=12838) | Placebo (N=12835)
Cardiac disorders (Cardiac disorders) | 35 | 13
Ear and labyrinth disorders (Ear and labyrinth disorders) | 3 | 1
Eye disorders (Eye disorders) | 48 | 27
Gastrointestinal disorders (Gastrointestinal disorders) | 1168 | 690
General disorders (General disorders) | 176 | 138
Investigations (Investigations) | 218 | 132
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 439 | 270
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 545 | 516
Nervous system disorders (Nervous system disorders) | 213 | 179
Psychiatric disorders (Psychiatric disorders) | 112 | 82
Renal and urinary disorders (Renal and urinary disorders) | 42 | 38
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 | 2
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 75 | 51
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1835 | 580
Vascular disorders (Vascular disorders) | 927 | 123 — Only non-serious adverse events considered by participant to be related to study treatment recorded

LIMITATIONS AND CAVEATS:
Participants may have SAEs reported in >1 category hence total participants affected across reported categories is less than total given.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No